CLINICAL TRIAL: NCT00170001
Title: Which Supraesophageal Reflux Symptoms Reliably Respond to PPI Therapy: A Large Simple Trial
Brief Title: Which Supraesophageal Reflux Symptoms Reliably Respond to Proton-Pump-Inhibitor (PPI) Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Yvonne Romero, Mayo Clinic Rochester, MN
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 452-05; IRUSESOM0376
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Gastroesophageal Reflux
Keywords: supraesophageal reflux; laryngopharyngeal symptoms; pharynx; esophagus
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar Pill
- Active Comparator (Active Comparator)
  Interventions: Drug: Nexium

INTERVENTIONS:
Drug: Nexium — 40 mg bid dosing
  Arms: Active Comparator
Drug: Sugar Pill — 40 mg BID
  Arms: Sugar pill

SUMMARY:
The investigators hypothesize that persons with the particular cluster of symptoms that are due to supraesophageal reflux (SER) will have complete resolution of those symptoms with adequate acid suppression when a PPI is administered for 6 months.

DETAILED DESCRIPTION:
Estimates suggest that up to 50% of Voice Clinic patients and 10% of ENT and Pulmonology outpatients seek medical care for chronic laryngopharyngeal symptoms resulting from supraesophageal reflux (SER). While many anecdotal and uncontrolled studies have shown significant clinical benefit with Proton Pump Inhibitors (PPIs), this conclusion has not been supported in small, randomized, placebo-controlled studies. The recent negative Vaezi trial (unpublished) was limited by bias introduced in the patient enrollment process due to reliance on physician diagnosis of SER. This bias became clear during conduction of the Supraesophageal Reflux Questionnaire (SRQ) Validation Study (Mayo, in press), which demonstrated that Otolaryngologists vary in their threshold for considering the diagnosis of SER. This project aims to remove selection bias from the study design.

Hypotheses/Questions: Our underlying assumptions are as follows: SER is due to the passage of gastric contents into the esophagus; and with adequate acid suppression provided by a PPI, there is less overall volume available to reflux, which should improve SER. We hypothesize that persons with the particular cluster of symptoms that are due to SER will have complete resolution of those symptoms with adequate acid suppression when PPI is administered for an adequate duration of time.

Primary Aim:

* To determine which symptom(s) (chronic cough, hoarseness, sore throat, globus sensation, or throat clearing) are completely ameliorated with PPI therapy and hence reflective of SER.

Secondary Aims:

* To determine which features of a patient's history are predictive of a positive response to PPI therapy, and which confer lack of response; and
* To develop a scoring system for the SRQ that would predict a diagnosis of SER.

Methods:

Design: Large simple randomized, double-blind, placebo-controlled trial of subjects with chronic laryngopharyngeal symptoms.

Population: Subjects will be recruited from Olmsted County and from General ENT Clinic and Pulmonary Chronic Cough Clinic.

Inclusion Criteria: Subjects must have at least 1 of 5 chronic (present for at least one month) and recurrent (at least twice per week) symptoms of interest.

Randomization: A dynamic allocation algorithm will be used by the Mayo Pharmacy to balance the treatment arms for confounding variables for treatment allocation.

Study Intervention: Either twice daily esomeprazole 40 mg or placebo for 6 months. Beyond a urine pregnancy test for women of child-bearing age, no other examination is required for enrollment or participation.

Follow-Up: Subjects will be contacted by phone monthly to assess symptoms, check compliance, and adverse events.

Primary Outcome: True responders will be those subjects who lack at least one of their initial symptoms by the 3-month time period, and remain asymptomatic at 4, 5 and 6 months.

Sample Size: Based on previous studies we anticipate a 30-40% placebo response rate at 3 months that will not be sustained at 6 months. We expect roughly 60% to completely respond to PPI therapy (i.e. 40% do not completely respond). Assuming 140 patients do not completely respond, we would need 350 patients on PPI therapy. Hence, 70 subjects will be randomized to receive PPI therapy and 30 randomized to placebo for each symptom group for a total N=500.

Analysis: Logistic regression.

Significance: This project will identify patients with laryngopharyngeal symptoms most likely to benefit from empiric PPI therapy. Until we have clarified which symptoms best respond and do not respond to therapy, we are bound to repeat the errors of the past. Finally, this project will further validate the SRQ for use in future trials.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint includes one of the following symptoms: chronic cough (dry, hacking, or nocturnal), hoarseness, sore throat, globus sensation, or throat clearing. These symptoms will be identified by a yes response to SRQ (Appendix 7) items 2, 3, 4, 5, 6, and 8. Furthermore, symptom(s) must be chronic (present for at least 1 month), and recurrent (at least twice per week). These criteria correspond to SRQ columns on page 3-5. The first column asks: When in your life did you first notice this symptom? A response with either number 2, 3, 4, or 5 meets criteria for chronic. The second column asks: How frequently have you noticed the symptom? A response with either number 3, 4, or 5 meets criteria for recurrent.

Exclusion Criteria:

* History of head and neck cancer/radiation/surgery (SRQ items 15, 16, 17)
* History of esophagus/stomach surgery (SRQ item 22)
* Peptic or duodenal ulcer disease; stomach or gastric ulcer disease; history of esophageal stricture, or Barrett's esophagus, or esophagitis, or tumor of the esophagus or stomach (SRQ item 23 and review of electronic surgical records of Mayo Clinic patients)
* Presence of alarm symptoms (hemoptysis, unexplained loss of 10 or more pounds in the past 3 months), obtained from Appendix 5 for Community Subjects, medical record for clinic subjects. History of dysphagia, defined as a yes answer to SRQ item 7.
* PPI use within 4 weeks, obtained from Appendix 5 for Community Subjects, medical record for clinic subjects
* Use of warfarin or digoxin, obtained from Appendix 5 for Community Subjects, medical record for clinic subjects
* Pregnancy at the time of enrollment, based on urine pregnancy test
* Inability to understand or read English at a 6th grade level
* Residence outside of the United States of America (USA)
* Age younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine which symptom(s) are predictive of SER based on a complete response to PPI therapy | 1 month

SECONDARY OUTCOMES:
To determine which symptoms demonstrate partial response with PPI therapy | 1 month
To determine which features of a patient's history are predictive of a positive response to PPI therapy | 1 month
To determine which features of a patient's history are predictive of a lack of response to PPI therapy | 1 month
To develop a scoring system for the Supraesophageal Reflux Questionnaire (SRQ) that would predict a diagnosis of SER | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Romero, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States